CLINICAL TRIAL: NCT02704169
Title: Comparing GTV Delineation With and Without Spatially Registered Endoscopy
Brief Title: Quantitative Endoscopy of H&N
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Princess Margaret Hospital, Canada (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UHN REB 13-5914-C
Record Dates: First submitted 2013-06-27; First posted 2016-03-09 (Estimated); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Head and Neck Cancer
Keywords: head and neck cancer; H&N cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Spatially registered endoscopy for H&N cancer (Experimental)
  Interventions: Other: Spatially registered endoscopy

INTERVENTIONS:
Other: Spatially registered endoscopy

SUMMARY:
The last decade has seen progressive advances in RT delivery, such as intensity modulated radiation therapy (IMRT)and image-guided radiation therapy (IGRT), which now allow highly precise radiation dose delivery. Together, IMRT and IGRT offer the potential of more selective treatment of the primary tumour and surrounding neck nodes by reducing the dose inflicted on critical organs at risk without compromising tumour dose and. IMRT has been shown to significantly decrease radiation-induced toxicity, and is now considered standard treatment for H&N tumors. With these advances in delivery technology, the accurate definition of the target is emerging as the weakest link in the radiotherapeutic treatment chain. Accurate target definition is the primary link on which all subsequent treatment planning and delivery depend and is therefore critical for successful RT. Incorrect target definition can result in poorer outcomes through either less tumour control, more normal tissue toxicity, or both. Computed x-ray tomography (CT) is the standard volumetric imaging modality for RT because of its high resolution, accurate definition of anatomy and its intrinsic measure of electron density necessary for accurate dose calculation. However, its ability to distinguish between tumour and normal tissue is limited due to a lack of contrast for structures of similar electron density and image artifacts for objects of high density. This additional noise can result in large inter-observation variability. Disease visible on endoscopy can be contoured and registered to the planning CT, allowing inclusion of superficial disease invisible on the volumetric CT image dataset into the treatment plan.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Histologic diagnosis of squamous cell carcinoma
* Primary cancer of the H&N
* Intention to treat using external beam radiation therapy as part of standard radiotherapy.
* Ability to provide written informed consent to participate in the study

Exclusion Criteria:

* Prior complete or partial radiation therapy to H&N
* Prior complete or partial surgery of the tumour
* Contraindications to full dose radiation therapy including pregnancy, lactation, connective tissue disorders, serious co-morbid illness
* Concurrent illness or condition that precludes subject from undergoing endoscopy or CT scanning
* Psychiatric or addictive disorders that preclude informed consent or adherence to protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-07; Primary Completion 2019-08-12 (Actual); Study Completion 2019-08-12 (Actual)

PRIMARY OUTCOMES:
Difference between endoscopic gross tumor volume contours (GTV-endo) and standard gross tumor volume contours (GTV-std) | 18 months
  Determine if spatially registered endoscopic gross tumor volume contours (GTV-endo) and standard gross tumor volume contours (GTV-std) are significantly different in primary H&N tumors treated with radiation therapy
Difference between inter-observer variation (V) of endoscopic gross tumor volume and of standard gross tumor volume | 18 months
  Determine if the inter-observer variation (V) of spatially registered endoscopic gross tumor volume contours is significantly less than standard gross tumor volume contours in primary H&N tumors treated with radiation therapy

SECONDARY OUTCOMES:
Difference between dose distribution using endoscopic gross tumor volume and using standard gross tumor volume | 18 months
  Determine if the dose distributions using spatially registered endoscopic GTV contours and standard GTV contours are significantly different in primary H&N tumors treated with radiation therapy with regard to both normal tissue radiation exposure and tumor coverage

CONTACTS AND LOCATIONS:
Overall Officials: John Cho, MD, Principal Investigator — The Princess Margaret Cancer Foundation
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Shi RB, Mirza S, Martinez D, Douglas C, Cho J, Irish JC, Jaffray DA, Weersink RA. Cost-function testing methodology for image-based registration of endoscopy to CT images in the head and neck. Phys Med Biol. 2020 Nov 13;65(20). doi: 10.1088/1361-6560/aba8b3. PMID 32702685